CLINICAL TRIAL: NCT03303248
Title: Evaluation of Web-based Transition Education to Enhance Transition Readiness and Health Service Utilization in Adolescents/Young Adults With Congenital Heart Disease
Brief Title: Evaluation of Web-based Transition Education to Enhance Transition Readiness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: University of Nebraska (Other)
Responsible Party: Principal Investigator, Karen Uzark, Clinical Professor of Cardiac Surgery and Pediatric Cardiology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HUM00130432
Record Dates: First submitted 2017-10-02; First posted 2017-10-05 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Congenital Heart Disease; Transition; Pediatric Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Web-based Educational Intervention (Experimental): This group of participants will be given access to a web-based educational resource in addition to the standard of care.
  Interventions: Behavioral: Web-based Educational Intervention
- Standard of Care (No Intervention): This group will be given only the standard of care during their clinic visit.

INTERVENTIONS:
Behavioral: Web-based Educational Intervention — A web-based educational tool, created for patients with congenital heart disease, will be given to patients using an ipad. This additional educational tool will be used with the standard of care visit with provider.
  Arms: Web-based Educational Intervention

SUMMARY:
The study looks to learn more about the helpfulness of web-based transition education and its effect on transition readiness and health service utilization in the adolescent and young adult congenital heart disease population.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with congenital heart disease
* Ages 13-25
* Routine outpatient cardiology follow-up visit

Exclusion Criteria:

* New patients to cardiology clinic
* Patients being evaluated for an acute medical problem
* Patients who do not speak English
* Severe neurocognitive impairment that precludes ability to complete the questionnaire

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change in transition readiness score, as measured by transition readiness survey | baseline, 12 months
  The transition readiness survey is used to measure a participant's self-reported knowledge about their health and readiness to take charge of their healthcare. Each item is scored from 1 to 5, where 1 means "No, I do not know how" and 5 means "Yes, I always do this when I need to." The overall score is determined by calculating the sum of all questions on a 100 point scale. A higher score indicates greater readiness for transition.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Uzark, PhD, CPNP, Principal Investigator — University of Michigan
Locations (1):
- C.S. Mott Children's Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Uzark K, Smith C, Donohue J, Yu S, Afton K, Norris M, Cotts T. Assessment of Transition Readiness in Adolescents and Young Adults with Heart Disease. J Pediatr. 2015 Dec;167(6):1233-8. doi: 10.1016/j.jpeds.2015.07.043. Epub 2015 Aug 19. PMID 26298627